CLINICAL TRIAL: NCT06873204
Title: RDA Cereal Fiber Clinical
Brief Title: Impact of Soluble Arabinoxylan and Rice Bran Fiber on the Gut Microbiome in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Rural Development Administration (RDA) of the Republic of Korea (Unknown)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-2024-881
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Gut microbiota; Dietary fiber; Soluble arabinoxylan; Rice bran fiber; Intestinal health; Butyrate-producing bacteria; Clostridium cluster IVa; Short-Chain Fatty Acids
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, double-blind, clinical trial (RCT).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Soluble Arabinoxylan (Experimental): Participants in this arm will receive soluble arabinoxylan for 3 consecutive weeks.
  Interventions: Dietary Supplement: Soluble Arabinoxylan
- Rice Bran (Experimental): Participants in this arm will consume rice bran fiber for 3 consecutive weeks.
  Interventions: Dietary Supplement: Rice Bran
- Maltodextrin (Placebo Comparator): Participants in this arm will consume maltodextrin for 3 consecutive weeks.
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Soluble Arabinoxylan — 10 grams of soluble arabinoxylan diluted in 200 mL of water, twice daily for 3 consecutive weeks.
  Arms: Soluble Arabinoxylan
Dietary Supplement: Rice Bran — 10 grams of rice bran fiber diluted in 200 mL of water, twice daily for 3 consecutive weeks.
  Arms: Rice Bran
Dietary Supplement: Maltodextrin (Placebo) — 10 grams of maltodextrin diluted in 200 mL of water, twice daily for 3 consecutive weeks.
  Arms: Maltodextrin

SUMMARY:
The importance of the gut microbiota for general health has been recently elucidated, but little is known about the impact of different types of nutrients on the gut microbiota. The soluble fiber in cereal by-products, arabinoxylan (AX), is known to be beneficial for generally promoting gut health. However, it is unclear whether consuming rice bran (RB), the source of AX, is equally helpful or better than consuming the extracted form of AX. This study aims to reveal the potential benefit of insoluble cereal bran fiber ingredients by comparing the effect of soluble arabinoxylan fiber alone and the mostly insoluble rice bran fiber, containing arabinoxylan, on intestinal health and gut microbiota. A placebo (maltodextrin) will be used as a control, with no significant changes expected in this group for the evaluated outcomes.

Participants will:

* Consume two different fiber supplements (soluble arabinoxylan or stabilized rice bran) as well as a placebo (maltodextrin) for 3 weeks each, separated by a 2-week washout period.
* Provide blood and stool samples at six different time points.
* Complete a food and gastrointestinal symptom diary during the intervention periods.

DETAILED DESCRIPTION:
Background:

This randomized, crossover clinical trial aims to evaluate the effects of two types of dietary fibers (soluble arabinoxylan and rice bran) compared to a control (maltodextrin) on gut microbiota and intestinal health in healthy adults aged 18-45. Insoluble rice bran, a fiber derived as a cereal by-product, may provide special support of a group of beneficial gut bacteria, and may compare well to its soluble arabinoxylan counterpart. This study will provide insights into whether rice bran, as a fiber source, offers additional benefits compared to the extracted soluble form alone.

Significance:

This study will contribute to the understanding of how different types of cereal fibers, specifically soluble arabinoxylan and rice bran, influence gut microbiota composition and overall intestinal health. The findings will have implications for dietary interventions aimed at promoting gut health, especially in relation to fiber intake from whole food sources compared to extracted fiber components.

Sample size:

25 subjects will be enrolled in the study to have a final number of at least 21, considering a 20% dropout rate.

The study involves three arms:

1. Soluble arabinoxylan: Participants will consume 10 grams of soluble arabinoxylan diluted in 200 mL of water, twice daily (morning and evening), for 3 weeks.
2. Rice bran: Participants will consume 10 grams of defatted, stabilized rice bran diluted in 200 mL of water, twice daily (morning and evening) for 3 weeks.
3. Maltodextrin: Participants will consume 10 grams of maltodextrin diluted in 200 mL of water, twice daily (morning and evening) for 3 weeks.

A two-week washout period will separate the three intervention phases to minimize carryover effects. The order in which participants receive the interventions will be randomized before the study starts.

Study Objectives:

The primary objective is to determine if rice bran fiber promotes the growth of Clostridium cluster IVa, a butyrate-producing bacterial group known to be beneficial for gut health. The secondary objective is to assess differences in the composition of gut microbiota and short-chain fatty acid production among the three interventions. Blood samples will be analyzed for barrier function proteins to further understand how each supplement influences gut integrity.

Study Procedures:

* Screening: Participants will undergo pre-screening via an online questionnaire and those who meet the criteria, will attend an in-person visit for physical measurements (height, weight, and BMI calculation) at the Clinical Research Center at Purdue University. A small amount of blood will be drawn for general health assessment.
* Interventions: Candidates who fully meet the inclusion criteria will be enrolled in the study. Once a week, they will stop at the Department of Food Science at Purdue University to receive sachets containing one of the three supplements described above. Participants will be instructed to consume one sachet in the morning and one in the evening, diluted in water. Each treatment will last for three weeks, followed by a two-week washout period.
* Sample Collection: Biological samples will be collected on the first and the last day of each intervention (days 1, 21, 35, 56, 70, and 91) and include stool and blood collection.
* The participants will be required to fill out a Diet History Questionnaire (DHQ) at the baseline (week 0) and at the end of the study (13th week) to evaluate whether changes in their dietary patterns occurred. 24-hour dietary recalls will also be administered at specific time points during the study to estimate nutrient intake (weeks 0, 1, 2, 3, 5, 6, 7,8, 10, 11, 12, and 13). Lastly, the short form of the International Physical Activity Questionnaire (IPAQ) will be applied at baseline (week 0) and the end of each treatment arm (weeks 3, 8, and 13) to evaluate the participants' physical activity patterns, as well as any eventual shifts throughout the study.
* Additionally, participants will be asked to complete a food and gastrointestinal symptom diary everyday during the intervention periods.

Data Analysis:

Gut microbiota composition will be assessed using DNA sequencing of stool samples, while blood samples will be analyzed for intestinal barrier function markers. Additionally, short-chain fatty acid concentrations in the stool will be measured to understand the metabolic effects of each fiber type on the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Men or women.
* Aged between 18-45 years.
* Body mass index between 18.5 and 25 kg/m².
* Able to read/speak English.

Exclusion Criteria:

* Gastrointestinal disorders (inflammatory bowel disease, irritable bowel syndrome, gluten sensitivity/intolerance, etc.).
* Those who took antibiotics 3 months before the study.
* Individuals taking regular medication or supplements that might affect the gut microbiota.
* Individuals undertaking weight-loss diets.
* Unstable body weight (±3 kg in the past 3 months), and individuals below 110 lb.
* Heavy drinkers (for men, consuming more than 4 drinks on any day or more than 14 drinks per week; for women, consuming more than 3 drinks on any day or more than 7 drinks per week).
* Smokers (those who have smoked 100 cigarettes in their lifetime and who currently smoke cigarettes, even every day or occasionally).
* Breastfeeding or pregnant women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of two test fibers (insoluble cereal bran and soluble arabinoxylan) and a control (maltodextrin) on gut beneficial bacteria | From enrollment to the end of treatment at 13 weeks.
  The primary outcome of the study is change in butyrogenic Clostridium cluster XIVa gut bacteria.

SECONDARY OUTCOMES:
Comparison of two tests (insoluble cereal bran and soluble arabinoxylan) and a control (maltodextrin) on fecal butyrate and intestinal barrier function | From enrollment to the end of treatment at 13 weeks.
  Secondary outcomes are fecal butyrate, gut barrier function protein (serum zonulin), and serum lipopolysaccharide-binding protein (LBP)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center at Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided